CLINICAL TRIAL: NCT02842710
Title: Staphylococcus Aureus Resistant to Methicillin (MRSA) Screening in Trauma
Acronym: TRAUMASARM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the study did not start due to a lack of staff
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/15/7856
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GeneXpert® (Experimental): Detection is carried out after a sample within the patient's nasal cavity. The swab containing the sample is placed in the PLC GeneXpert® Cepheid . The analysis takes one hour . The results leave automatically.
  Interventions: Device: GeneXpert®

INTERVENTIONS:
Device: GeneXpert® — Detection is carried out after a sample within the patient's nasal cavity. The swab containing the sample is placed in the PLC GeneXpert® Cepheid . The analysis takes one hour . The results leave automatically.

SUMMARY:
The main objective of this study and to know the incidence of healthy carriers of Staphylococcus aureus resistant méti- patients supported for fracture of the proximal femur .

This assessment will be made preoperatively by a nasal sampling and analysis through it by rapid Polymerase Chain Reaction method GeneXpert® .

DETAILED DESCRIPTION:
There are 85,000 fractures of the upper extremity in France each year. This is a frequent pathology in fragile patients. The characteristics in terms of comorbidities, age, sex and survival are well known from the literature. While secondary mechanical complications to surgery, hovering around 6 to 8%, mortality at one year is very high (around 25%).

Postoperative infection after a fracture of the upper end of the femur ranges from 2 to 8% depending on the series. This complication is responsible for morbidity and excess mortality linked to the need for revision surgery, prolongation of hospitalization and antibiotic treatment.

In elective surgery, detection of Staphylococcus aureus resistant to methicillin is systematic and recommended in many countries, preoperative level of the nasal cavity. Parvizi then Goya believe that this port increased from four to nine times the occurrence of infection at the surgical site.

Various epidemiological studies have shown the presence of Staphylococcus aureus in over 30% of patients. This prevalence is lower in the French population. An estimated 70% the proportion of Staphylococcus aureus in the periprosthetic infections, and 30% related specifically to the methicillin-resistant Staphylococcus aureus.

Today there is no consensus on what to have vis-à-vis the detection of a hand and the other hand treatment of patients.

The healthy carrier in the population overtake admitted to the trauma unit is unclear.

It is therefore necessary to know these effects among patients with multiple pathologies.

For methods of detection, the usual system and directed by swabbing and cultured with 90% sensitivity specificity of 100%. The demoyens existence of early detection as GeneXpert® Cepheid® lets get this result is in an hour with a specificity of 98% and a sensitivity of 100%.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated in the trauma unit for fractures of the proximal femur belong to a social security scheme patient

Exclusion Criteria:

* Minor patient
* Presence of abrasions
* MRSA history
* Open fracture
* Ongoing infectious process
* Patients under judicial protection , guardianship
* Pregnant or breastfeeding women
* patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06-04 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of Staphylococcus aureus resistant to methicillin nasal carriage in the population supported to trauma emergencies | 12 months
  To evaluate the prevalence of Staphylococcus aureus resistant to methicillin nasal carriage in the population supported to trauma emergencies

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Reina, Dr, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No